CLINICAL TRIAL: NCT01193790
Title: Evaluation of Coblation Channeling in Treating Chronic Tonsillitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: I. Braverman, MD, Hillel Yaffe MC, Hadera, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43-2001
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Tonsillitis
Keywords: chronic tonsillitis; radio-frequency coblation; radio-frequency coblation in chronic tonsillitis treatment
MeSH Terms: conditions — Tonsillitis

ARMS (1):
- Coblation (Experimental)
  Interventions: Procedure: Coblation channeling

INTERVENTIONS:
Procedure: Coblation channeling — The combination of the energy and the fluid creates a "plasma" field containing highly ionized particles (coblation). The ionized particles have sufficient energy to break organic molecular bonds that can remove tissue selectively without excessive heat production and subsequent damage to the surrounding tissue. Treatment of the tonsillar crypts and tissue by coblation may decrease antigen and immune system interaction and inflammation.

SUMMARY:
The investigators wish to evaluate coblation channeling in the treatment of chronic tonsillitis.

DETAILED DESCRIPTION:
The tonsillar crypts play an important role in chronic tonsillitis. They are covered by stratified epithelium and may be initiated via the epithelium to mount immune responses to various presenting antigens. Go M. et al, investigated the expression and function of tight junctions in the epithelium of human palatine tonsils from patients with tonsillar hypertrophy or recurrent tonsillitis. These studies suggested unique expression of tight junctions in human palatine tonsillar epithelium, and it was suggested that the crypt epithelium may possess an epithelial barrier different from that of the surface epithelium.

Bacteria within biofilms are resistant to host defenses and antibiotics. The presence of bacterial biofilms within the tissue and crypts of inflamed tonsils may explain the chronicity and recurrent characteristics of some forms of tonsillitis. There is strong anatomical evidence for the presence of bacterial biofilms in chronically diseased tonsils.

Our hypothesis was that treatment of the crypts and tonsillar tissue may decrease the possible antigen-immune system interaction and inflammation.

The combination of the radio frequency energy and the fluid creates a "plasma" field containing highly ionized particles. The ionized particles have sufficient energy to break organic molecular bonds that can remove tissue selectively without excessive heat production and damage the surrounding tissue. Employing this new technique, the investigators will try to eliminate the cause for chronic tonsillitis.

The combination of the radio frequency energy and the fluid creates a "plasma" field containing highly ionized particles. The ionized particles have sufficient energy to break organic molecular bonds that can remove tissue selectively without excessive heat production and damage the surrounding tissue. Employing this new technique, the investigators will try to eliminate the cause for chronic tonsillitis.

Our hypothesis was that treatment of the crypts and tonsillar tissue may decrease the possible antigen-immune system interaction and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* suffering from at least 4 episodes of tonsillitis in past year.
* suffering from recurrent or chronic sore throat.
* suffering from irregular tonsils with crypts, slight redness or enlargement.

Exclusion Criteria:

* suffering from mouth ulcers or other oral מחלת ריריות
* allergic to the type of medication included in the study.
* suffering from gastrointestinal (GI) reflux or chronic הפרשה הוסטנזלית
* contraindication to medical or surgical treatment.
* suffering from peritonsillar abscess.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
RF coblation may be promising in treating chronic tonsillitis. | 2 years

SECONDARY OUTCOMES:
RF coblation reduces tonsillar volume and pain in comparison to surgery; may be performed as an out-patient procedure. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe MC,, Hadera, Israel